CLINICAL TRIAL: NCT05372562
Title: Risk Factors for the Recurrent Postoperative Macular Edema Treated With OZURDEX
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Chun Zhang, professor, Peking University
Other Study IDs: IRB00006761-M2022205
Record Dates: First submitted 2022-04-22; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with recurrent macular edema: after intravitreal injection of OZURDEX, patients with macular edema relapse during follow-up were recruited.
- patients without recurrent edema: after intravitreal injection of OZURDEX, patients without macular edema relapse during follow-up were recruited.

SUMMARY:
Patients who were diagnosed as postoperative CME and administrated with intravitreal OZURDEX injection were reviewed. Outcome will include best-corrected visual acuity (BCVA), intraocular pressure (IOP) and central macular thickness (CMT). Recurrent CME and corresponding treatments were recorded.

DETAILED DESCRIPTION:
Patients who were diagnosed as postoperative CME after uneventful intraocular surgery and administrated with intravitreal OZURDEX injection were reviewed. All patients underwent ophthalmic examinations at the initial visit and were followed up at months 1, 2, 3 and 6 with measurement of best-corrected visual acuity (BCVA), intraocular pressure (IOP) and central macular thickness (CMT). Recurrent CME and corresponding treatments were recorded. Risk factors of recurrent CME were analyzed

ELIGIBILITY:
Inclusion Criteria:

* patients who were diagnosed as postoperative CME after successful phacoemulsification or vitrectomy and administrated with intravitreal dexamethasone implant (OZURDEX, Allergan, Inc, California, USA) injection were reviewed.

Exclusion Criteria:

* patients with retinal vascular diseases, including retinal vein occlusion (RVO), diabetic retinopathy (DR), hypertensive retinopathy, retinal artery occlusion (RAO), Coats disease, Eales disease;
* patients with macular disease before surgery, such as age-related macular degeneration (ARMD), macular choroidal neovascularization (CNV), myopic macular degeneration, macular hole (MH), epiretinal membrane(ERM);
* patients with uveitis before surgery, including anterior, intermediate, posterior and generalized uveitis;
* patients with autoimmune disease, such as ankylosing spondylitis (AS), Vogt-Koyanagi-Harada (VKH) disease, Behcet disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who were diagnosed as postoperative CME after successful phacoemulsification or vitrectomy and administrated with intravitreal dexamethasone implant (OZURDEX, Allergan, Inc, California, USA) injection
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | All patients underwent the examination at baseline and changes were followed up at months 1, 2, 3 and 6.
  Measurement of best-corrected visual acuity (BCVA) by Snellen scale and was converted into logarithmic scale (LogMAR).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hosipital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided